CLINICAL TRIAL: NCT03443466
Title: A Comparative Study of Success Rate, Efficacy, Safety Between Electric Stimulation-guided Epidural Catheter Placement and the Loss of Resistance Conventional Method for Cesarean Section
Brief Title: Efficacy and Safety of Electric Stimulation-guided Epidural Anesthesia for Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Sewoon Medical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Sang Sik Choi, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015GR0703 (RegionalStimⓇ)
Record Dates: First submitted 2018-01-30; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Epidural Anesthesia
Keywords: Electric stimulation; Cesarean section

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural electrical stimulation (EES) (Experimental): n=20
  Interventions: Device: Epidural electrical stimulation (EES)
- Loss of resistance (LOR) (Active Comparator): n=20
  Interventions: Device: Loss of resistance (LOR)

INTERVENTIONS:
Device: Epidural electrical stimulation (EES) — Using loss of resistance technique and electrical stimulation
  Arms: Epidural electrical stimulation (EES)
Device: Loss of resistance (LOR) — Using loss of resistance technique only
  Arms: Loss of resistance (LOR)

SUMMARY:
Forty pregnant women (36 to 41 weeks gestation) will randomly allocate to two groups. Groups will be defined based on the method used to identify the epidural space for epidural anesthesia: the loss of resistance group (n=20) and the epidural electric stimulation group (n=20). Pain during the cesarean section will be assessed using a numerical visual analog scale and maternal satisfaction by a post-partum interview. The success rate of epidural anesthesia, maternal satisfaction, and neonatal Apgar scores will be compared between groups.

DETAILED DESCRIPTION:
Investigators will place epidural catheter in the epidural space using loss of resistance technique, and will confirm correct placement of the epidural catheter using electric stimulation.

Epidural catheter placement, electric stimulation, and confirmation of response is followed:

Patients will be placed in the left lateral decubitus position. The site will be aseptically prepared and 1% lidocaine will be infiltrated to the skin. An 18-gauge Tuohy needle will be inserted midline of L4/5 interspinous space.

For the LOR group, after identification of the epidural space, the Tuohy needle will be stopped, and a 20-gauge epidural catheter will be advanced through the Touhy needle.

The same process will be followed for the EES group. In addition, the epidural space will be confirmed by epidural electric stimulation using a 20-gauge epidural catheter (RegionalStimTm, Sewoon Medical Co., Ltd, Seoul, Korea, 800 mm) with a conductive guidewire (conductive guidewire, Nitinol, 1100 mm).

After confirming there is no reverse flow of cerebrospinal fluid or blood with aspiration, 3 mL of 1% lidocaine, with 15 mcg of epinephrine (1:200000), will be injected through the epidural catheter as test dose. If there is no response to the test dose, patients will be moved to the operating room. In operating room, 20 mL of 2% lidocaine, 2 mL of bicarbonate (total volume 22 mL) will be administered in divided doses.

Blood pressure (BP), heart rate (HR), oxygen saturation (SpO2), and neurologic assessment findings will be monitored.

Pain relief in cesarean section is assessed in the visual analogue scale (VAS) score. A 10 point VAS, where 0 is no pain and 10 is unbearable pain, is used to assess pain during labor. The scale is assessed after epidural anesthesia. Differences in the VAS we used to assess the efficacy of the epidural anesthesia in decreasing labor pain. Comparison of the change in VAS between groups is used to compare pain control of the two methods. The success of epidural anesthesia is defined by sensory block, without motor block, and a decrease in pain score after adequate dosing of epidural medication. Failure of epidural anesthesia is defined in several ways. Objective outcome include conversion to general anesthesia, conversion to any different form of anesthesia, or pain during surgery.

Patient satisfaction will be evaluated by a postpartum interview. Satisfaction is graded between a score of 1-5, where 1 represent very unsatisfied and 5 represent very satisfied. Patients will indicate a score of 1 to 5.

One- and 5-minute Apgar scores will be compared to assess the effect of epidural electric stimulation on the neonate. Additional time required for epidural electric stimulation will be determined by the difference (in seconds) from LOR to identification of the epidural space through electric stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were at 36 to 41 weeks' gestation and admitted in labor to the university clinic for cesarean section were included. Patients were American Society of Anesthesiologists (ASA) physical status of I or II, and were scheduled to receive epidural anesthesia.

Exclusion Criteria:

* Skin infection at the injection site
* Difficult catheter placement owing to previous lumbar spinal surgery or deformity
* Presence of a hemostatic disorder or use of antiplatelet therapy
* Presence of a cardiac pacemaker.
* Removal of patient

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Maternal
Enrollment: 40 (Estimated)
Dates: Start 2015-03-11 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Success rate of epidural anesthesia | Up to 6 months
  Evaluation parameter : Accuracy comparison between loss of resistance and epidural electrical stimulation

SECONDARY OUTCOMES:
Maternal satisfaction | Up to 6 months
  Patient satisfaction will be evaluated by a postpartum interview. Satisfaction was graded by patients from 1 to 5, where 1 represented very unsatisfied and 5 represented very satisfied
Neonatal Apgar score | Up to 6 months
  The neonatal apgar scores from 0 to 10 were measured at 1 and 5 minutes to assess the effect of electrical stimulation on the fetus; Scores 7 and above are generally normal, 4 to 6 fairly low, and 3 and below are generally regarded as critically low
Procedure-related complications | Up to 6 months
  The number of times dural puncture or intravascular insertion was performed by Tuohy needle of epidural catheter during epidural anesthesia
Minimum electrical current to elicit a response in the epidural electrical stimulation group | Up to 6 months
  Minimum current stimulus to confirm that the epidural catheter is located in the epidural space between 0 and 5mA ;mA (frequency, 1 Hz; pulse width, 300 ms)
Additional time for epidural electrical stimulation | Up to 6 months
  * Determined by the difference (in seconds) from loss of resistance(LOR) to identification of the epidural space through electrical stimulation
  * Measure : seconds (from observation of LOR to confirmation of the epidural space by electric stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Sik Choi, MD, PhD, Principal Investigator — Korea University Guro Hiospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva M, Halpern SH. Epidural analgesia for labor: Current techniques. Local Reg Anesth. 2010;3:143-53. doi: 10.2147/LRA.S10237. Epub 2010 Dec 8. PMID 23144567
- [Background] Wantman A, Hancox N, Howell PR. Techniques for identifying the epidural space: a survey of practice amongst anaesthetists in the UK. Anaesthesia. 2006 Apr;61(4):370-5. doi: 10.1111/j.1365-2044.2006.04534.x. PMID 16548958
- [Background] Eappen S, Blinn A, Segal S. Incidence of epidural catheter replacement in parturients: a retrospective chart review. Int J Obstet Anesth. 1998 Oct;7(4):220-5. doi: 10.1016/s0959-289x(98)80042-3. PMID 15321183
- [Background] Hermanides J, Hollmann MW, Stevens MF, Lirk P. Failed epidural: causes and management. Br J Anaesth. 2012 Aug;109(2):144-54. doi: 10.1093/bja/aes214. Epub 2012 Jun 26. PMID 22735301
- [Background] Tsui BC, Tarkkila P, Gupta S, Kearney R. Confirmation of caudal needle placement using nerve stimulation. Anesthesiology. 1999 Aug;91(2):374-8. doi: 10.1097/00000542-199908000-00010. PMID 10443599
- [Background] Tsui BC, Gupta S, Finucane B. Confirmation of epidural catheter placement using nerve stimulation. Can J Anaesth. 1998 Jul;45(7):640-4. doi: 10.1007/BF03012093. PMID 9717595
- [Derived] Kim YS, Kim HS, Jeong H, Lee CH, Lee MK, Choi SS. Efficacy of electrical stimulation on epidural anesthesia for cesarean section: a randomized controlled trial. BMC Anesthesiol. 2020 Jun 10;20(1):146. doi: 10.1186/s12871-020-01063-1. PMID 32522156